CLINICAL TRIAL: NCT01900236
Title: Integrating ENGagement and Adherence Goals Upon Entry iENGAGE to Control HIV
Acronym: iENGAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of North Carolina (Other); University of Washington (Other); Johns Hopkins University (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Michael J Mugavero, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1R01AI103661 (NIH)
Record Dates: First submitted 2013-07-02; First posted 2013-07-16 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: HIV
Keywords: Patients newly initiating outpatient HIV medical care
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Control arm participants will receive standard clinical care (i.e. receive usual clinic treatment)
- Motivation Behavioral Technique (Experimental): Behavioral: 4 sessions of tailored, interactive agenda based on behavioral motivational interviewing (MI) techniques. Each iENGAGE intervention session includes: interventionist-delivered educational content for managing HIV medical care appointment-keeping and information sessions for learning to manage HIV medications. The goal of this intervention is for the participant to establish early behaviors that help him/her to arrive at scheduled medical appointments and learn to take medications as prescribed during the initial year of HIV care in order in order to achieve viral suppression and improve overall health.
  Interventions: Behavioral: Based on behavioral motivational interviewing (MI) technique

INTERVENTIONS:
Behavioral: Based on behavioral motivational interviewing (MI) technique — In addition to receiving standard clinic care, the intervention will have a tailored, interactive agenda for each of the 4 sessions based on behavioral motivational interviewing (MI) technique. The goal of this intervention is for the participant to establish early behaviors that help him/her to arrive at scheduled medical appointments and learn to take medications as prescribed during the initial year of HIV care in order to in order to achieve viral suppression and improve overall health.
  Arms: Motivation Behavioral Technique

SUMMARY:
iENGAGE is a 4 session, in-clinic behavioral intervention that is delivered to new clinic patients during the first year of HIV care on a flexible delivery schedule, with intervention visits scheduled to coincide with HIV medical care visits. Interventionists from each participating collaborating site will be trained centrally to implement the iENGAGE protocol. Following study enrollment and baseline assessment, participants will be randomized to treatment as usual and intervention groups. For intervention-arm participants, each iENGAGE intervention session includes: interventionist-delivered educational content for managing HIV medical care appointment-keeping and information sessions for learning to manage HIV medications. The intervention will have a tailored, interactive agenda for each of the 4 sessions based on behavioral motivational interviewing (MI) techniques. The goal of this intervention is for the participant to establish early behaviors that help him/her to arrive at scheduled medical appointments and learn to take medications as prescribed during the initial year of HIV care in order to improve overall health.

DETAILED DESCRIPTION:
The Centers for Disease Control's Retention In Care (CDC RIC) and the Participating and Communicating Together (PACT) antiretroviral therapy (ART) adherence interventions have shown success in the literature, and they are well suited to target the two essential HIV adherence behaviors needed to achieve better overall health: HIV medical visit adherence and ART adherence. While these original interventions target each of these behaviors separately, the comprehensive iENGAGE intervention combines these two approaches to address the experience of an individual who is initiating HIV care. Upon entry to care, knowledge, motivation, and skills for adherence to HIV medical visits and ART must be learned rapidly. Jointly targeting these behaviors offers a distinct advantage over addressing them separately.

iENGAGE integrates CDC RIC and PACT through their common intervention targets with the assistance of trained interventionists, who will maintain contact with the new patient to educate and assist with reinforcing the importance of adherence to care. While the actions required to attend HIV medical care appointments and take medications properly are distinct, each is influenced by an individual's personal motivation and skills for self-management of HIV infection and overall health; these principles are the focus of the intervention sessions for this protocol .

During this intervention, our team will make every effort to protect all participants' confidential and private information in order to minimize possible study-associated risks. In addition, the follow up measurement plan for this study is unique, as it aims to utilize the X060831001: Unsolicited R24 for the Centers for AIDS Research (CFAR) Network of Integrated Clinical Sciences, (CNICS), PI Michael Saag) secure electronic data infrastructure, which has existing defined protocols for the protection of human subjects data, including a data management core that is housed at the collaborating site at the University of Washington.

Stigma Supplement (Michael J. Mugavero, Janet M. Turan, Bulent Turan)

As part of this supplement, the research team has incorporated multi-item questionnaire measures of stigma into baseline and final data collection for the iENGAGE trial. The goal of Aim 1 is to examine the longitudinal associations and potential causal mechanisms in the relationships between dimensions of HIV-related stigma and HIV visit adherence, antiretroviral therapy (ART) adherence, and viral load suppression, among control participants in the study. In addition, in Aim 2, we will examine the effects of the iENGAGE intervention on dimensions of stigma, by comparing changes in stigma in the two arms of the Randomized Controlled Trial (RCT).

For Aim 3, after participants have completed the 48-week iENGAGE intervention, we will conduct up to 40 individual in-depth face-to-face qualitative interviews with selected participants using a separate informed consent process. Topics to be explored in these interviews include qualitative exploration of how HIV-related stigma and other intersectional stigmas affect engagement in HIV care, as wells as exploring how participation in the iENGAGE intervention may have influenced the participant's experiences of anticipated, internalized, and experienced stigma; as well as disclosure concerns and actual disclosure behavior.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* Newly establishing HIV care at study site
* Age 18 years or older
* English speaking

Exclusion Criteria:

* Not willing or able to provide informed consent
* Received prior outpatient HIV care
* Completed >1 primary care visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2013-12; Primary Completion 2017-06-30 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Viral load (VL) suppression (<200c/ml) among patients newly initiating outpatient HIV medical care | 48 weeks
  VL suppression is defined as <200 copies/ml of blood

SECONDARY OUTCOMES:
Viremia Copy Years (VCY) | 96 weeks
  VCY is the area under the curve estimate of cumulative VL burden
Visit adherence | First provider visit to 48 weeks and 96 weeks
  We will calculate visit adherence as a proportion that captures the number of "attended" visits in the numerator and the number of total scheduled visits ("attended" plus "no show") in the denominator during study period.
4 month visit constancy | First provider visit to 48 weeks and 96 weeks
  We will evaluate visit constancy as the proportion of pre-specified time intervals with at least 1 attended clinic visit during the study period. We will use 4 month time interval
Time to viral load (VL) suppression | First provider visit to first VL suppression with administrative censoring at 12 months
  We will calculate time to VL suppression (defined as <200 copies/ml) as the time in days from the first medical provider visit to the first date with VL suppression. Kaplan-Meier analyses and Cox proportional hazards analyses will be used to generate survival curves and to estimate the median time to VL suppression.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Mugavero, MD, Principal Investigator — University of Alabama at Birmingham
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The Johns Hopkins HIV Care Program, Baltimore, Maryland
  - UNC Infectious Diseases Clinic, Chapel Hill, North Carolina
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Yigit I, Modi RA, Weiser SD, Johnson MO, Mugavero MJ, Turan JM, Turan B. Effects of an intervention on internalized HIV-related stigma for individuals newly entering HIV care. AIDS. 2020 Sep 1;34 Suppl 1(Suppl 1):S73-S82. doi: 10.1097/QAD.0000000000002566. PMID 32881796
- [Derived] Shaw S, Modi R, Mugavero M, Golin C, Quinlivan EB, Smith LR, Roytburd K, Crane H, Keruly J, Zinski A, Amico KR. HIV Standard of Care for ART Adherence and Retention in Care Among HIV Medical Care Providers Across Four CNICS Clinics in the US. AIDS Behav. 2019 Apr;23(4):947-956. doi: 10.1007/s10461-018-2320-1. PMID 30377981
- [Derived] Modi RA, Mugavero MJ, Amico RK, Keruly J, Quinlivan EB, Crane HM, Guzman A, Zinski A, Montue S, Roytburd K, Church A, Willig JH. A Web-Based Data Collection Platform for Multisite Randomized Behavioral Intervention Trials: Development, Key Software Features, and Results of a User Survey. JMIR Res Protoc. 2017 Jun 16;6(6):e115. doi: 10.2196/resprot.6768. PMID 28623185